CLINICAL TRIAL: NCT00763113
Title: A Prospective Randomized Study on Vanguard Cruciate Retaining Versus Vanguard High Flex Posterior Stabilized Total Knee System in the Early Range of Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMET CA 01
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Vanguard PS Knee
  Interventions: Device: Vanguard PS Knee
- 2 (Active Comparator): Vanguard CR Knee
  Interventions: Device: Vanguard CR Knee

INTERVENTIONS:
Device: Vanguard PS Knee — Vanguard PS Knee
  Arms: 1
Device: Vanguard CR Knee — Vanguard CR Knee
  Arms: 2

SUMMARY:
Main Objectives are: Test Difference in terms of early ROM between Vanguard FB CR and Vanguard FB PS. Knees; Demonstrate the comparable ROM of high flex PS to CR.

ELIGIBILITY:
Patients need total knee replacement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2007-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Knee Society Score | 6weeks, 6months, 1 year

SECONDARY OUTCOMES:
WOMAC | 6weeks, 6months, 1 year
Oxford Knee | 6weeks, 6months, 1 year
Complication | Anytime

CONTACTS AND LOCATIONS:
Overall Officials: David Martin, MD, Principal Investigator — St. Catharines Hospital
Locations (1):
- St. Catharines Hospital, Ontario, Canada